CLINICAL TRIAL: NCT06538025
Title: Post-stroke Fatigue and Its Correlation With Family Functioning in Patients With First-episode Stroke
Brief Title: Correlation Between Family Functioning and PSF
Status: Completed | Type: Observational
Sponsor: Meichun Shu (Other)
Responsible Party: Sponsor-Investigator, Meichun Shu, Principal Investigator, First Affiliated Hospital of Wenzhou Medical University
Organization: First Affiliated Hospital of Wenzhou Medical University (Other)
Other Study IDs: Meichun Shu
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Stroke
Keywords: post-stroke fatigue; family functioning
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the present study, the investigators investigate the effect of family functioning on PSF in neurologic stroke patients in the early stages of the disease by surveying the current status of post-stroke fatigue to provide theoretical support for clinical care.

ELIGIBILITY:
Inclusion Criteria:

* patients whose clinical manifestations met the diagnostic criteria for stroke and whose stroke was confirmed by imaging (cranial computed tomography or cranial magnetic resonance imaging)
* those with first-episode stroke and in a stable condition
* those who were conscious and able to cooperate with the investigation
* those who gave informed consent and volunteered to participate in the study

Exclusion Criteria:

* patients with severe aphasia
* those with severe cognitive impairment who were unable to cooperate with examinations or questionnaires
* those with malignant tumours
* those with degenerative diseases of the central nervous system, such as Parkinson's disease
* those who were unable to cooperate with the doctor in the examination for other reasons
* those with a previous history of mental illness
* those with other recent major stressful life events, such as divorce or death of a loved one
* those with pre-stroke fatigue (PrSF)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with first-episode stroke admitted to the Department of Neurology of our hospital between October 2021 and July 2022 were rigorously screened using convenience sampling.
Sampling Method: Non-Probability Sample
Enrollment: 212 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
activities of daily living | Before hospitalization
  modified Barthel index (MBI) is a tool most commonly used to assess the ability of stroke patients to perform activities of daily living. The measurement consists of 10 items, namely feeding, bed-to-wheelchair transfer, personal hygiene, toileting, bathing, walking, walking up and down stairs, dressing and bowel control, with a total score of 100. The lower the MBI score is, the more severe the dysfunction and the greater the dependence. The degree of dependence was categorised into four grades, with ≤40 points categorised as severe dependence (all items required care from others - poor), 41-60 points categorised as moderate dependence (most items required care from others - fair) and 61-90 points and 90-100 points, categorised as mild or no dependence, respectively (few or no items required care from others - good).
family adaptation, partnership, growth, affection and resolve (APGAR) score | First day after hospitalization
  assess patients' satisfaction with family functioning. It was developed to measure the five dimensions of adaptation, partnership, growth, affection and resolve in five separate questions. Each question was assigned a score of 0-2, with a total score of 0-10 points. The degree of family dysfunction was divided based on the total score, with 7-10 points defined as good family function, 4-6 points as moderate family dysfunction and 0-3 points as severe family dysfunction, with a Cronbach's α coefficient of 0.94
Post-stroke fatigue | Day 5 of hospitalization
  Post-stroke fatigue was scored using the Fatigue Severity Scale, which is mainly designed to assess the severity of physical and mental fatigue felt by patients as a result of the disease. When assessing stroke patients using the FSS, some scholars have diagnosed a score of ≥36 points as indicative of PSF. The FSS is comprised of a total of nine entries, each of which is scored on a 7-point Likert scale ranging from 1 to 7. A score of 1 indicates a 'strongly disagree' response to the corresponding entry, and a score of 7 represents a 'strongly agree' response to the corresponding entry. The final FSS score for the patient was obtained by summing the total score of the nine entries. The higher the score is, the more severe the patient's fatigue。
Sleep Disturbances | Day 5 of hospitalization
  The Athens Insomnia Scale (AIS) is used to measure the sleep quality of patients during the study period. AIS is an internationally recognized self-assessment scale for sleep quality, consisting of 8 items. The scale is a 4-point Likert scale, scored 0, 1, 2, or 3, with 0 representing "not at all" and 3 representing a "severe" impact. The total score is 24 points. Scores ranging from 0-4 indicate no sleep disturbances, 4-6 suggest possible insomnia, and scores above 6 represent insomnia. The higher the score, the poorer the sleep quality and the more severe the sleep problems. The Cronbach's alpha coefficient for this scale is 0.875.
Anxiety and Depression | Day 5 of hospitalization
  The Hospital Anxiety and Depression Scale (HADS) is composed of 14 items divided into two subscales: the depression subscale (7 items) and the anxiety subscale (7 items). Scores from 0 to 7 indicate no symptoms, 8 to 10 suggest possible symptoms, and 11 to 21 indicate definite symptoms. The overall Cronbach's alpha coefficient for the scale, as well as those of the anxiety and depression subscales, are 0.88 and 0.81, respectively.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Meichun Shu, Wenzhou, Zhejiang
  - Xianchai Hong, Wenzhou, Zhejiang